CLINICAL TRIAL: NCT04287023
Title: Effects of Physical Therapy on Gait Parameters in Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Viorela Mihaela Ciortea, MD, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversitateaMFHCluj
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Physical therapy (Experimental): 1 physical therapists and groups of 10 patients during the sessions
  Interventions: Other: group physical therapy
- Individual physical therapy (Active Comparator): 1 physical therapist and 1 patient during the sessions
  Interventions: Other: individual physical therapy

INTERVENTIONS:
Other: individual physical therapy — cardiovascular warm-up activities, stretching exercises, strengthening exercises, functional, gait and balance training, recreational games and ended with relaxation exercises - individual
  Arms: Individual physical therapy
Other: group physical therapy — cardiovascular warm-up activities, stretching exercises, strengthening exercises, functional, gait and balance training, recreational games and ended with relaxation exercises - groups of 10 patients
  Arms: Group Physical therapy

SUMMARY:
Parkinson disease is a progressive neurologic disorder characterized by motor impairments which alter the walking capacity, and lead to reduced walking speed, decreased stride length and increased double support time. Physical therapy interventions are an important part of the non-pharmacological treatment for Parkinson disease. The purpose of this study is to assess whether there is a different outcome regarding improvement of gait parameters, when applying a physical therapy program in an individual or in a group manner.

The study setting is the Clinical Rehabilitation Hospital in Cluj-Napoca, Cluj county, Romania. Patients will be randomly divided into 2 groups, and were prescribed either individual (1 patient and 1 physical therapist) or group physical therapy (6 patients and 1 physical therapist). Treatment protocol includes 10 sessions of physical therapy, in the same room setting and performed the same routine of exercises, except for the 3 breaks during the sessions in the group therapy for informal socialization. Walking speed will be measured by two validated instruments, the 6-minute walk test and the 10-meter walk test, before and after treatment.

DETAILED DESCRIPTION:
The rehabilitation protocol for the individual physical therapy will consist of cardiovascular warm-up activities, stretching exercises, strengthening exercises, functional, gait and balance training, recreational games and ended with relaxation exercises. In addition, the group protocol will follow the exact same pattern, except for 5-10 minute breaks for informal socialization between participants, at the beginning of the session, mid-session and at the end of the session.

Also, both groups will have access to external cues, which will be applied during a variety of tasks and environmental situations, like gait initiation and termination, heel strike and push-off, sideways and backwards stepping, walking while dual tasking, and walking over various surfaces and long distances.

All patients will be evaluated at the beginning and at the end of the physical therapy program. The evaluation includes the 6-minute walking test and the 10-meter walking test. Gait speed for each participant will be calculated as the ratio between the walked distance and the time unit, and it was measured in meters/seconds.

ELIGIBILITY:
Inclusion Criteria:

* stable medication usage;
* Hoehn and Yahr stage 2, 3 or 4;
* ability to walk independently or by using an assistive walking device;
* no severe cognitive impairments (Mini-Mental State Examination - MMSE score, ≥24);
* no other severe neurologic, cardiopulmonary or orthopedic disorders;
* not having participated in a PT or rehabilitation program in the previous 2 months.

Exclusion Criteria:

* not stable medication usage;
* Hoehn and Yahr stage 1;
* inability to walk independently or by using an assistive walking device;
* severe cognitive impairments (Mini-Mental State Examination - MMSE score, below 24);
* other severe neurologic, cardiopulmonary or orthopedic disorders;
* having participated in a PT or rehabilitation program in the previous 2 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Change in walking speed | at baseline and after 10 days
  meters/seconds - the 6 minute walk test and 10 meter walk test

CONTACTS AND LOCATIONS:
Overall Officials: Viorela Ciortea, Principal Investigator — Rehabilitation Hospital Cluj-Napoca
Locations (1):
- Rehabilitation Hospital, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No
upon request